CLINICAL TRIAL: NCT06916611
Title: Heart Failure With Preserved Ejection Fraction and Its Cardiac MR Characteristics of Different Subtypes
Status: Active, not recruiting | Type: Observational
Sponsor: The Affiliated Hospital of Xuzhou Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: XYFY2023-KL187-01
Record Dates: First submitted 2025-01-20; First posted 2025-04-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: HFpEF; Heart Failure With Preserved Ejection Fraction
Keywords: Heart Failure with Preserved Ejection Fraction，HFpEF; Cardiac Magnetic Resonance Imaging，CMR

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients diagnosed with HFpEF: Diagnostic criteria for HFpEF:
  * Age = 50 years old ② Cardiac color ultrasound EF 50% ③ Symptoms / signs of heart failure and increased natriuretic peptide levels during hospitalization / visit (BNP 100 pg/mL or NT-proBNP 400 pg / mL).
  Interventions: Other: Cardiac Magnetic Resonance Imaging

INTERVENTIONS:
Other: Cardiac Magnetic Resonance Imaging — This study included patients who were diagnosed with HFpEF and had completed CMR.

SUMMARY:
Using cardiac magnetic resonance imaging technology, the ejection fraction of heart failure (HFpEF) and different subtypes of cardiac magnetic resonance characteristics, and combined with the clinical characteristics and prognosis of the patient, explore the value of cardiac magnetic resonance in disease diagnosis, classification, treatment and prognosis, and provide new ideas for clinical practice.

DETAILED DESCRIPTION:
1. Study Objectives To compare clinical characteristics among HFpEF patients with different comorbidity subtypes (hypertension, type 2 diabetes, renal insufficiency, obesity).

   To identify distinct cardiac magnetic resonance (CMR) features associated with HFpEF and its comorbidity subtypes.

   To evaluate prognostic differences (mortality, heart failure readmission, healthcare costs) across HFpEF subtypes.
2. Study Design Type: Single-center, prospective, observational cohort study. Duration: April 1, 2023 - December 31, 2026. Sample Size: 500 HFpEF patients, with ~200 patients per subgroup.
3. Data Collection Framework

   Baseline Data:

   Clinical Parameters:

   Demographics (age, gender, BMI). Comorbidities (hypertension, diabetes, renal function). Biochemical markers (BNP/NT-proBNP, HbA1c, lipid profile, renal function). Medications (ACE inhibitors, beta-blockers, diuretics).

   Imaging Data:

   Echocardiography: Left ventricular ejection fraction (LVEF ≥50%). CMR: Ventricular volumes, mass, strain analysis, T1 mapping, and late gadolinium enhancement (LGE).

   Follow-Up Protocol:

   Frequency: Every 6 months post-discharge.

   Endpoints:

   Primary: Cardiovascular mortality, HF-related readmission. Secondary: Changes in CMR parameters, medication adjustments, healthcare utilization.
4. Subgroup Classification

   Comorbidity Subgroups:

   HFpEF + Hypertension. HFpEF + Type 2 Diabetes. HFpEF + Renal Insufficiency. HFpEF + Obesity. Control Group: HFpEF patients without the above comorbidities.
5. CMR Protocol

   Imaging Sequences:

   Cine imaging for ventricular function. T1 mapping for myocardial fibrosis assessment. LGE for scar detection. Post-Processing: Analysis of myocardial strain, extracellular volume (ECV), and perfusion reserve.
6. Statistical Analysis

   Methods:

   Regression analysis for associations between CMR features and clinical outcomes.

   Survival analysis (Kaplan-Meier, Cox proportional hazards models). Subgroup comparisons using ANOVA or non-parametric tests. Software: SPSS 20.0 (significance threshold: p <0.05).
7. Ethical and Data Management Privacy Protection: De-identified data storage with restricted access. Data Validation: Double-entry verification for 10% of randomly selected cases. Compliance: Adherence to institutional review board (IRB) guidelines and GCP standards.

ELIGIBILITY:
Inclusion Criteria:

* Age is 50 years old.
* Cardiac color ultrasound shows an ejection fraction (EF) of 50% or more.
* Symptoms / signs of heart failure and increased natriuretic peptide levels during hospitalization / visit (BNP 100 pg/mL or NT-proBNP 400 pg / mL).

Exclusion Criteria:

* Severe liver and kidney insufficiency
* Severe valvular heart disease (severe, severe severe) or known infiltrative or hypertrophic cardiomyopathy
* Malignant tumors and severe hematological diseases
* severe infection
* Autoimmune system diseases

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In the patients who were diagnosed with "cardiac insufficiency / heart failure" from April 1,2023 to December 31,2026, the medical records were retrieved and the enrolled patients were determined according to the enrollment criteria and the exclusion criteria.
  Subgroup selection: ① HFpEF combined with hypertension
  * HFpEF is complicated with type 2 diabetes mellitus ③ HFpEF combined with renal insufficiency ④ HFpEF combined with obesity Control group: ①HFpEF patients
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of Cardiovascular death | follow - up every 6 months; up to 24 - months
Rate of readmission of heart failure | follow - up every 6 months; up to 24 - months

SECONDARY OUTCOMES:
Body Temperature | Baseline
  Measure body temperature every morning on an empty stomach using an electronic thermometer, with the unit being degrees Celsius (℃)
Blood Glucose Levels | Baseline
  Draw blood on an empty stomach in the morning and detect fasting blood glucose using a biochemical analyzer, with the unit being mmol/L; measure 2 - hour post - prandial blood glucose using a portable blood glucose meter, with the unit being mmol/L.
Brain Natriuretic Peptide (BNP) | Baseline
  Detect BNP levels using an electrochemiluminescence immunoassay analyzer, with the unit being picograms per milliliter (pg/mL).
Glycated Hemoglobin (HbA1c) | Baseline
  Detect glycated hemoglobin using high - performance liquid chromatography, and the result is expressed as a percentage (%).
Blood Pressure | Baseline
  Measure blood pressure once in the morning and once in the evening every day using a blood pressure monitor, with the unit being millimeters of mercury (mmHg)
Heart Rate | Baseline
  Continuously monitor the heart rate using an electrocardiogram monitor, with the unit being beats per minute (bpm).

CONTACTS AND LOCATIONS:
Locations (1):
- the Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No
Considering the patient's privacy and the next steps in our research program